CLINICAL TRIAL: NCT02515253
Title: A Randomised Control Trial of an Individual Bra Prescription Versus Standard Care for Women With Larger Breasts and Breast Pain
Brief Title: A Breast Support Intervention for Women With Breast Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Emma Burnett, PhD Research Student, University of Portsmouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BP-01
Record Dates: First submitted 2015-07-27; First posted 2015-08-04 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Mastodynia
Keywords: Breast Pain; Mastalgia; Bras; Breast Support
MeSH Terms: conditions — Mastodynia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prescription group (Experimental): Participants in this group will receive the standard care for benign breast pain sufferers (administered by the Queen Alexandra Hospital in Portsmouth) and will also attend the Department of Sport and Exercise Science at the University of Portsmouth for an individual bra prescription. Participants will be prescribed an appropriate bra to wear over an eight week intervention period.
  Interventions: Other: Bra prescription; Other: Standard Care
- Standard care group (Other): Participants in this group will receive the standard care for benign breast pain sufferers administered by the Queen Alexandra Hospital in Portsmouth.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Bra prescription
  Arms: Prescription group
Other: Standard Care

SUMMARY:
The purpose of this study is to assess whether prescribing a bra to participants results in an improvement in the Patient Global Impression of Change (PGIC) compared to participants who receive standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 years of age and above.
* Experiencing breast pain of any severity.
* Participants must be able to speak and read English fluently
* Participants must be a resident within the local area and not planning to move out of the area within the study timeline
* Participant must have attended the Queen Alexandra (QA) hospital for an assessment of their breast pain.
* Participant is willing and able to give informed consent for participation in the study.
* Participant is self-reported to be between a 34 and 40 under band size and a DD to G bra cup size.
* Able to walk on a treadmill for up to two minutes unaided and be able to walk unaided up and down a small set of steps (assessed verbally by the clinicians at QA hospital)
* Participants must be able to comply with the study procedures

Exclusion Criteria:

* Participants are receiving any additional treatment for their breast pain that is not part of standard care (recommendation for a bra fit, topical ibuprofen, breast pain leaflet) including any cancer treatment
* Participants have had any surgery to the breasts within the last year
* Participants are currently pregnant or have been pregnant or breast fed in the past year
* Planning to undertake any activities or lifestyle changes which may affect their levels of breast pain e.g. trying for a baby, changing oral contraceptive, having breast surgery.
* Participant's data will be excluded from the analysis if they do not complete either survey at four or eight weeks (at least one follow up survey needs to be completed).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Burnett, MRes, Principal Investigator — University of Portsmouth; Joanna Scurr, PhD, Study Chair — University of Portsmouth
Locations (2):
- United Kingdom (2):
  - Department of Sport and Exercise Science, University of Portsmouth, Portsmouth
  - Breast Care Services, Queen Alexandra Hospital, Portsmouth

RESULTS

PARTICIPANT FLOW:
Groups:
- Prescription Group: Participants in this group will receive the standard care for benign breast pain sufferers (administered by the Queen Alexandra Hospital in Portsmouth) and will also attend the Department of Sport and Exercise Science at the University of Portsmouth for an individual bra prescription. Participants will be prescribed an appropriate bra to wear over an eight week intervention period.
  Bra prescription
  Standard Care
- Standard Care Group: Participants in this group will receive the standard care for benign breast pain sufferers administered by the Queen Alexandra Hospital in Portsmouth.
  Standard Care
Period: Overall Study
Arm/Group | Prescription Group | Standard Care Group
Started | 17 | 16
Completed | 10 | 8
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prescription Group | Standard Care Group | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9) | 32 (6) | 39 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Breast Pain [Median (Standard Deviation); unit: scores on a scale] — Numerical rating scale 0 = No pain 10 = Worst possible pain
  scores on a scale | 6 (2) | 2 (2) | 6 (2)
Quality of Life (Physical Component Summary) [Mean (Standard Deviation); unit: scores on a scale] — 0-100 scale 0 = maximum effect on the physical component of quality of life 100 = no effect on the physical component of quality of life
  scores on a scale | 49.3 (7.4) | 55.0 (5.7) | 51.8 (7.1)
Quality of Life (Mental Component Summary) [Mean (Standard Deviation); unit: MCS score] — 0-100 scale 0 = maximum effect on mental component of quality of life 100 = no effect on mental component of quality of life
  MCS score | 45.6 (9.6) | 44.8 (8.8) | 45.2 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Impression of Change (PGIC)
Description: Participants will complete the PGIC as part of a questionnaire four weeks after receiving their treatment for benign breast pain
  1. = Very much improved (better outcome)
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse (worse outcome)
Time Frame: four weeks post intervention
Population: Percentage of those who scored "Very much improved" or "much improved" in each group
Measure: Number; unit: percentage of VMI/MI respondents
Arm/Group | Prescription Group | Standard Care Group
Number analyzed (Participants) | 9 | 8
percentage of VMI/MI respondents | 55 | 25

2. Primary Outcome: Patient Global Impression of Change (PGIC)
Description: Participants will complete the PGIC as part of a questionnaire eight weeks after receiving their treatment for benign breast pain
Time Frame: eight weeks post intervention
Population: Percentage of those scoring "very much improved" or "much improved"
Measure: Number; unit: percentage
Arm/Group | Prescription Group | Standard Care Group
Number analyzed (Participants) | 10 | 8
percentage | 50 | 25

ADVERSE EVENTS:
Arm/Group | Prescription Group | Standard Care Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes